CLINICAL TRIAL: NCT03437759
Title: Mesenchymal Stem Cells Derived Exosomes Promote Healing of Large and Refractory Macular Holes
Brief Title: MSC-Exos Promote Healing of MHs
Acronym: MSCs
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin Medical University (Other)
Responsible Party: Principal Investigator, Xiaomin Zhang, Principal Investigator, Tianjin Medical University Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015KY-05
Record Dates: First submitted 2018-01-23; First posted 2018-02-19 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Macular Holes
Keywords: macular hole (MH); exosomes; mesenchymal stem cells; pars plana vitrectomy
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Our intervention is to add treatment of exosomes derived from mesenchymal stem cells (MSC-Exo) after pars plana vitrectomy(PPV) and ILM peeling.
  Interventions: Biological: exosomes derived from mesenchymal stem cells (MSC-Exo)
- Control group (No Intervention): Control group that receives treatment of only pars plana vitrectomy(PPV) and ILM peeling.

INTERVENTIONS:
Biological: exosomes derived from mesenchymal stem cells (MSC-Exo) — After air-liquid exchange, 50μg or 20μg MSC-Exo in 10μl PBS was dripped into vitreous cavity around MH, leaving 20% SF6 or air as tamponade .
  Arms: Experimental group

SUMMARY:
Purpose: To assess the safety and efficacy of mesenchymal stem cells (MSCs) and MSC-derived exosomes (MSC-Exos) for promoting healing of large and refractory macular holes (MHs).

Hypothesis: MSC and MSC-Exo therapy may promote functional and anatomic recovery from MH. MSC-Exo therapy may be a useful and safe method for improving visual outcomes of surgery for refractory MHs.

DETAILED DESCRIPTION:
Based on the purpose and hypothesis,the participants with large and longstanding idiopathic MHs underwent vitrectomy, internal limiting membrane peeling, MSC or MSC-Exo intravitreal injection, and heavy silicon oil, air, 20% SF6, or 14% C3F8 tamponade. MSCs were isolated from human umbilical cord, and MSC-Exos were isolated from supernatants of MSCs via sequential ultracentrifugation. At the time of study enrollment, as well as physical examinations, best-corrected visual acuity (BCVA) and intraocular pressure will be measured and fundoscopy be performed. All diagnoses of MH are going to confirmed via spectral-domain optical coherence tomography (OCT), and the minimum linear diameter (MLD) of each MH will be measured parallel to the retinal pigment epithelium.The participants are going to be followed up for at least 6 months via BCVA measurement, fundoscopy, OCT, and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

1.Clinical diagnosis of idiopathic macular hole whose diameter is greater than 400 microns

Exclusion Criteria:

1. Only one functional eye
2. In other clinical trials.
3. Other diseases which can affect visual acuity, such as cataract, diabetic retinopathy, glaucoma, corneal diseases, etc.
4. Eye had undergone vitrectomy or scleral buckling, cataract surgery, Nd:YAG laser less than one month ago.
5. Contralateral eye has poor prognosis than the study eye.
6. Idiopathic or autoimmune uveitis history.
7. Aphakic eye
8. Physical condition is poor that can not keep prone position.
9. Secondary macular lesions
10. The equivalent spherical diopter of the study eye before any refractive correction or cataract surgery, which is greater than 6.0d or above 26mm of the ocular axis of the study eye.
11. Intraocular pressure is higher than 25mmHg
12. Within ocular inflammation, such as eye blepharitis, scleritis, keratitis and conjunctivitis.
13. Systemic condition is poor, such as the poor control of diabetes and hypertension, myocardial infarction, cerebrovascular accident, renal failure and so on,and the researchers assessed those who are unable to complete the trail.

Max Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Macular holes closure | baseline to 24 weeks post-surgery
  Minimum linear diameter (MLD) of the hole measured by OCT

SECONDARY OUTCOMES:
Best corrected visual acuity(BCVA) | baseline to 24 weeks post-surgery
  BCVA using a Landolt C acuity chart method

CONTACTS AND LOCATIONS:
Overall Officials: Rong X Li, MD,PhD, Principal Investigator — Tianjin Medical University Eye Hospital
Locations (1):
- Tianjin Medical University Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rahmani B, Tielsch JM, Katz J, Gottsch J, Quigley H, Javitt J, Sommer A. The cause-specific prevalence of visual impairment in an urban population. The Baltimore Eye Survey. Ophthalmology. 1996 Nov;103(11):1721-6. doi: 10.1016/s0161-6420(96)30435-1. PMID 8942862
- [Result] Kelly NE, Wendel RT. Vitreous surgery for idiopathic macular holes. Results of a pilot study. Arch Ophthalmol. 1991 May;109(5):654-9. doi: 10.1001/archopht.1991.01080050068031. PMID 2025167
- [Result] Michalewska Z, Michalewski J, Cisiecki S, Adelman R, Nawrocki J. Correlation between foveal structure and visual outcome following macular hole surgery: a spectral optical coherence tomography study. Graefes Arch Clin Exp Ophthalmol. 2008 Jun;246(6):823-30. doi: 10.1007/s00417-007-0764-5. Epub 2008 Apr 2. PMID 18386040
- [Result] Ezra E, Gregor ZJ; Morfields Macular Hole Study Ggroup Report No. 1. Surgery for idiopathic full-thickness macular hole: two-year results of a randomized clinical trial comparing natural history, vitrectomy, and vitrectomy plus autologous serum: Morfields Macular Hole Study Group RAeport no. 1. Arch Ophthalmol. 2004 Feb;122(2):224-36. doi: 10.1001/archopht.122.2.224. PMID 14769600
- [Result] Suda K, Hangai M, Yoshimura N. Axial length and outcomes of macular hole surgery assessed by spectral-domain optical coherence tomography. Am J Ophthalmol. 2011 Jan;151(1):118-127.e1. doi: 10.1016/j.ajo.2010.07.007. PMID 20970769
- [Result] Del Priore LV, Kaplan HJ, Bonham RD. Laser photocoagulation and fluid-gas exchange for recurrent macular hole. Retina. 1994;14(4):381-2. doi: 10.1097/00006982-199414040-00018. No abstract available. PMID 7817035
- [Result] Johnson RN, McDonald HR, Schatz H, Ai E. Outpatient postoperative fluid-gas exchange after early failed vitrectomy surgery for macular hole. Ophthalmology. 1997 Dec;104(12):2009-13. doi: 10.1016/s0161-6420(97)30064-5. PMID 9400759
- [Result] Ohana E, Blumenkranz MS. Treatment of reopened macular hole after vitrectomy by laser and outpatient fluid-gas exchange. Ophthalmology. 1998 Aug;105(8):1398-403. doi: 10.1016/S0161-6420(98)98019-8. PMID 9709749
- [Result] Liggett PE, Skolik DS, Horio B, Saito Y, Alfaro V, Mieler W. Human autologous serum for the treatment of full-thickness macular holes. A preliminary study. Ophthalmology. 1995 Jul;102(7):1071-6. doi: 10.1016/s0161-6420(95)30909-8. PMID 9121755
- [Result] Wells JA, Gregor ZJ. Surgical treatment of full-thickness macular holes using autologous serum. Eye (Lond). 1996;10 ( Pt 5):593-9. doi: 10.1038/eye.1996.136. PMID 8977788
- [Result] Kim JY, Kwon OW. VITRECTOMY FOR REFRACTORY MACULAR HOLE. Retin Cases Brief Rep. 2015 Fall;9(4):265-8. doi: 10.1097/ICB.0000000000000183. PMID 26398430
- [Result] Kozy DW, Maberley AL. Closure of persistent macular holes with human recombinant transforming growth factor-beta 2. Can J Ophthalmol. 1996 Jun;31(4):179-82. PMID 8804755
- [Result] Rizzo S, Belting C, Genovesi-Ebert F, Cresti F, Vento A, Martini R. Successful treatment of persistent macular holes using "heavy silicone oil" as intraocular tamponade. Retina. 2006 Oct;26(8):905-8. doi: 10.1097/01.iae.0000250006.76155.3d. PMID 17031291
- [Result] Cillino S, Cillino G, Ferraro LL, Casuccio A. TREATMENT OF PERSISTENTLY OPEN MACULAR HOLES WITH HEAVY SILICONE OIL (DENSIRON 68) VERSUS C2F6. A PROSPECTIVE RANDOMIZED STUDY. Retina. 2016 Apr;36(4):688-94. doi: 10.1097/IAE.0000000000000781. PMID 26418444
- [Result] Michalewska Z, Michalewski J, Adelman RA, Nawrocki J. Inverted internal limiting membrane flap technique for large macular holes. Ophthalmology. 2010 Oct;117(10):2018-25. doi: 10.1016/j.ophtha.2010.02.011. Epub 2010 Jun 11. PMID 20541263
- [Result] Morizane Y, Shiraga F, Kimura S, Hosokawa M, Shiode Y, Kawata T, Hosogi M, Shirakata Y, Okanouchi T. Autologous transplantation of the internal limiting membrane for refractory macular holes. Am J Ophthalmol. 2014 Apr;157(4):861-869.e1. doi: 10.1016/j.ajo.2013.12.028. Epub 2014 Jan 10. PMID 24418265
- [Result] De Novelli FJ, Preti RC, Ribeiro Monteiro ML, Pelayes DE, Junqueira Nobrega M, Takahashi WY. Autologous Internal Limiting Membrane Fragment Transplantation for Large, Chronic, and Refractory Macular Holes. Ophthalmic Res. 2015;55(1):45-52. doi: 10.1159/000440767. Epub 2015 Nov 17. PMID 26569390
- [Result] Jiang Y, Zhang Y, Zhang L, Wang M, Zhang X, Li X. Therapeutic effect of bone marrow mesenchymal stem cells on laser-induced retinal injury in mice. Int J Mol Sci. 2014 May 27;15(6):9372-85. doi: 10.3390/ijms15069372. PMID 24871366
- [Result] Yu B, Shao H, Su C, Jiang Y, Chen X, Bai L, Zhang Y, Li Q, Zhang X, Li X. Exosomes derived from MSCs ameliorate retinal laser injury partially by inhibition of MCP-1. Sci Rep. 2016 Sep 30;6:34562. doi: 10.1038/srep34562. PMID 27686625
- [Result] Zhang L, Zheng H, Shao H, Nian H, Zhang Y, Bai L, Su C, Liu X, Dong L, Li X, Zhang X. Long-term therapeutic effects of mesenchymal stem cells compared to dexamethasone on recurrent experimental autoimmune uveitis of rats. Invest Ophthalmol Vis Sci. 2014 Aug 14;55(9):5561-71. doi: 10.1167/iovs.14-14788. PMID 25125599
- [Result] Chen X, Shao H, Zhi Y, Xiao Q, Su C, Dong L, Liu X, Li X, Zhang X. CD73 Pathway Contributes to the Immunosuppressive Ability of Mesenchymal Stem Cells in Intraocular Autoimmune Responses. Stem Cells Dev. 2016 Feb 15;25(4):337-46. doi: 10.1089/scd.2015.0227. Epub 2016 Jan 29. PMID 26650818
- [Result] Li G, Yuan L, Ren X, Nian H, Zhang L, Han ZC, Li X, Zhang X. The effect of mesenchymal stem cells on dynamic changes of T cell subsets in experimental autoimmune uveoretinitis. Clin Exp Immunol. 2013 Jul;173(1):28-37. doi: 10.1111/cei.12080. PMID 23607419
- [Result] Zhang X, Ren X, Li G, Jiao C, Zhang L, Zhao S, Wang J, Han ZC, Li X. Mesenchymal stem cells ameliorate experimental autoimmune uveoretinitis by comprehensive modulation of systemic autoimmunity. Invest Ophthalmol Vis Sci. 2011 May 16;52(6):3143-52. doi: 10.1167/iovs.10-6334. PMID 21296818
- [Result] Machalinska A, Kawa M, Pius-Sadowska E, Stepniewski J, Nowak W, Roginska D, Kaczynska K, Baumert B, Wiszniewska B, Jozkowicz A, Dulak J, Machalinski B. Long-term neuroprotective effects of NT-4-engineered mesenchymal stem cells injected intravitreally in a mouse model of acute retinal injury. Invest Ophthalmol Vis Sci. 2013 Dec 23;54(13):8292-305. doi: 10.1167/iovs.13-12221. PMID 24265016
- [Result] Rotenstreich Y, Tzameret A, Kalish SE, Belkin M, Meir A, Treves AJ, Naglera A, Sher I. [A novel system for minimally invasive transplantation of bone marrow derived stem cells as a thin layer in the subretina and extravascular spaces of the choroid--for treatment of retinal degeneration]. Harefuah. 2015 Feb;154(2):84-8, 138. Hebrew. PMID 25856858
- [Result] Yu B, Zhang X, Li X. Exosomes derived from mesenchymal stem cells. Int J Mol Sci. 2014 Mar 7;15(3):4142-57. doi: 10.3390/ijms15034142. PMID 24608926
- [Result] Doeppner TR, Herz J, Gorgens A, Schlechter J, Ludwig AK, Radtke S, de Miroschedji K, Horn PA, Giebel B, Hermann DM. Extracellular Vesicles Improve Post-Stroke Neuroregeneration and Prevent Postischemic Immunosuppression. Stem Cells Transl Med. 2015 Oct;4(10):1131-43. doi: 10.5966/sctm.2015-0078. Epub 2015 Sep 3. PMID 26339036
- [Result] Xin H, Li Y, Liu Z, Wang X, Shang X, Cui Y, Zhang ZG, Chopp M. MiR-133b promotes neural plasticity and functional recovery after treatment of stroke with multipotent mesenchymal stromal cells in rats via transfer of exosome-enriched extracellular particles. Stem Cells. 2013 Dec;31(12):2737-46. doi: 10.1002/stem.1409. PMID 23630198
- [Result] Katakowski M, Buller B, Zheng X, Lu Y, Rogers T, Osobamiro O, Shu W, Jiang F, Chopp M. Exosomes from marrow stromal cells expressing miR-146b inhibit glioma growth. Cancer Lett. 2013 Jul 10;335(1):201-4. doi: 10.1016/j.canlet.2013.02.019. Epub 2013 Feb 16. PMID 23419525
- [Result] Xin H, Li Y, Buller B, Katakowski M, Zhang Y, Wang X, Shang X, Zhang ZG, Chopp M. Exosome-mediated transfer of miR-133b from multipotent mesenchymal stromal cells to neural cells contributes to neurite outgrowth. Stem Cells. 2012 Jul;30(7):1556-64. doi: 10.1002/stem.1129. PMID 22605481
- [Result] Maltman DJ, Hardy SA, Przyborski SA. Role of mesenchymal stem cells in neurogenesis and nervous system repair. Neurochem Int. 2011 Sep;59(3):347-56. doi: 10.1016/j.neuint.2011.06.008. Epub 2011 Jun 21. PMID 21718735
- [Result] Joyce N, Annett G, Wirthlin L, Olson S, Bauer G, Nolta JA. Mesenchymal stem cells for the treatment of neurodegenerative disease. Regen Med. 2010 Nov;5(6):933-46. doi: 10.2217/rme.10.72. PMID 21082892
- [Result] Singh MS, Balmer J, Barnard AR, Aslam SA, Moralli D, Green CM, Barnea-Cramer A, Duncan I, MacLaren RE. Transplanted photoreceptor precursors transfer proteins to host photoreceptors by a mechanism of cytoplasmic fusion. Nat Commun. 2016 Nov 30;7:13537. doi: 10.1038/ncomms13537. PMID 27901042
- [Result] Pearson RA, Gonzalez-Cordero A, West EL, Ribeiro JR, Aghaizu N, Goh D, Sampson RD, Georgiadis A, Waldron PV, Duran Y, Naeem A, Kloc M, Cristante E, Kruczek K, Warre-Cornish K, Sowden JC, Smith AJ, Ali RR. Donor and host photoreceptors engage in material transfer following transplantation of post-mitotic photoreceptor precursors. Nat Commun. 2016 Oct 4;7:13029. doi: 10.1038/ncomms13029. PMID 27701378
- [Result] Yeo RW, Lai RC, Zhang B, Tan SS, Yin Y, Teh BJ, Lim SK. Mesenchymal stem cell: an efficient mass producer of exosomes for drug delivery. Adv Drug Deliv Rev. 2013 Mar;65(3):336-41. doi: 10.1016/j.addr.2012.07.001. Epub 2012 Jul 7. PMID 22780955
- [Result] Bai L, Shao H, Wang H, Zhang Z, Su C, Dong L, Yu B, Chen X, Li X, Zhang X. Effects of Mesenchymal Stem Cell-Derived Exosomes on Experimental Autoimmune Uveitis. Sci Rep. 2017 Jun 28;7(1):4323. doi: 10.1038/s41598-017-04559-y. PMID 28659587
- [Result] Hillenkamp J, Kraus J, Framme C, Jackson TL, Roider J, Gabel VP, Sachs HG. Retreatment of full-thickness macular hole: predictive value of optical coherence tomography. Br J Ophthalmol. 2007 Nov;91(11):1445-9. doi: 10.1136/bjo.2007.115642. Epub 2007 May 2. PMID 17475704
- [Result] Xin H, Li Y, Chopp M. Exosomes/miRNAs as mediating cell-based therapy of stroke. Front Cell Neurosci. 2014 Nov 10;8:377. doi: 10.3389/fncel.2014.00377. eCollection 2014. PMID 25426026